CLINICAL TRIAL: NCT03931915
Title: Phase III Clinical Study to Evaluate Efficacy and Safety of TAK-385 40 mg Compared With Leuprorelin in Patients With Endometriosis
Brief Title: Clinical Study to Evaluate Efficacy and Safety of TAK-385 40 mg Compared With Leuprorelin in Patients With Endometriosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ASKA Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TAK-385/3-A
Record Dates: First submitted 2019-04-24; First posted 2019-04-30 (Actual); Last update posted 2020-12-11 (Actual); Status verified 2020-07

CONDITIONS: Endometriosis
MeSH Terms: conditions — Endometriosis | interventions — relugolix; Leuprolide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TAK-385 (Experimental): TAK-385 40 mg administered orally once daily before breakfast + Leuprorelin placebo administered subcutaneously once every 4 weeks
  Interventions: Drug: TAK-385
- Leuprorelin acetate (Active Comparator): TAK-385 placebo administered orally once daily before breakfast + Leuprorelin acetate 1.88 mg / 3.75 mg administered subcutaneously once every 4 weeks
  Interventions: Drug: Leuprorelin acetate

INTERVENTIONS:
Drug: TAK-385 — TAK-385 40 mg tablets + Leuprorelin acetate placebo injection
  Other Names: relugolix
  Arms: TAK-385
Drug: Leuprorelin acetate — TAK-385 placebo tablets + Leuprorelin acetate 1.88 mg / 3.75 mg injection
  Arms: Leuprorelin acetate

SUMMARY:
The objective is to evaluate the efficacy and safety of TAK-385 40 mg orally administrated once daily for 24 weeks compared with Leuprorelin [once/4 weeks, 3.75 or 1.88 mg subcutaneously (SC)/time] in patients with endometriosis.

DETAILED DESCRIPTION:
This study is a phase III, multicenter, randomized, double-blind, parallel-group study to investigate the efficacy and safety of TAK-385 40 mg once daily compared with leuprorelin (once/4 weeks, 3.75 or 1.88 mg SC/time) in premenopausal subjects ≥ 20 years of age with endometriosis. 320 women with endometriosis will be enrolled in the study. This study consists of screening of approximately 1 to 6 weeks, run-in of approximately 3 to 6 weeks, treatment of 24 weeks, and follow-up of 4 weeks. After signing the informed consent form, subjects should record their symptoms in the electronic patient diary every day. During run-in period, daily data will be collected in the electronic patient diary for calculation of the baseline values for the efficacy evaluation.Following run-in period, subjects will receive investigational products (TAK-385 + leuprorelin placebo or TAK-385 placebo + leuprorelin) under double blind. During this study, subjects will visit the study center to undergo the designated examinations and evaluations at each visit. Safety will be assessed throughout the study by monitoring adverse events, vital signs, physical examinations, clinical laboratory tests, 12-lead electrocardiograms (ECG), and assessments of bone mineral density.Subjects will visit the study center to undergo the designated examinations and evaluations at 28 days after final administration.

ELIGIBILITY:
Inclusion Criteria:

1. The participant is a premenopausal Japanese woman aged 20 years or older at the time consent is obtained.
2. The participant with endometriosis that falls under one of the following. However, in case of recurrence after surgery, it must be diagnosed again by either of the following.

   * The participant who has been diagnosed with endometriosis by Laparotomy or Laparoscopy.
   * The participant who has been confirmed ovarian chocolate cyst by Magnetic Resonance Imaging (MRI) or ultrasonic examination (vaginal, transabdominal or rectal).
   * The participant who has been diagnosed with clinical endometriosis and has the symptom of either induration of Douglas cavum, restriction of uterine mobility or pelvic tenderness confirmed by internal or rectal examination.
3. The participant must have dysmenorrhea or pelvic pain associated with endometriosis, of which either 1 or both should be at least "moderate" as determined by the investigator or subinvestigator using the B&B scale.
4. The participant must have maximum VAS score > 30 for pelvic pain associated with endometriosis.
5. The participant has experienced regular menstrual cycles (25 to 38 days) that should include menstrual bleeding of at least 3 consecutive days (at least 3 regular menstrual cycles to be confirmed).
6. The participant agrees to use routinely adequate contraception from signing of informed consent throughout the duration of the study.

Exclusion Criteria:

1. The participant has the following drug usage:

   * Use of the following drugs within 24 weeks:bisphosphonate preparation or other investigational agent
   * Use of the following drugs within 16 weeks (for 1-, 3- and 6-month sustained-release preparations, within 20, 28 and 40 weeks, respectively): gonadotropin-releasing hormone (GnRH) analogues, danazol, or aromatase inhibitors.
   * Use of the following drugs within 8 weeks:dienogest, oral contraceptive or sex hormone preparations (norethindrone, norethisterone, medroxyprogesterone, estrogen, or other progestins, etc.)
   * Use of the following drugs (excluding drugs for external use and supplements) within 4 weeks :anti-coagulant drugs, anti-platelet drugs, tranexamic acid, selective estrogen receptor modulators, activated vitamin D preparations, other vitamin D preparations, calcitonin, ipriflavone, steroid hormones, vitamin K preparations, teriparatide, or denosumab
2. The participant has received TAK-385 (including placebo) in a previous clinical study.
3. The participant has ovarian chocolate cyst of 10 cm or more and over 40 years old at the time imaging test is performed.
4. The participant has a history of panhysterectomy or bilateral oophorectomy.
5. The participant has had markedly abnormal uterine bleeding or anovulatory bleeding, as determined by the investigator or subinvestigator.
6. The participant has nondiagnosable abnormal genital bleeding.
7. The participant has a current history of thyroid gland disorder with irregular menstruation, or has a potential for irregular menstruation due to thyroid gland disorder, as determined by the investigator or subinvestigator.
8. The participant has uterine fibroid requiring treatment.
9. The participant has lower abdominal pain due to irritable bowel syndrome or severe interstitial cystitis.
10. The participant has a previous or current history of pelvic inflammatory disease within 8 weeks.
11. The participant has a previous or current history of osteoporosis, osteopenia, or other metabolic bone diseases.
12. The participant has a positive cervical cytology result [other than Negative for Intraepithelial Lesion or Malignancy (NILM) in accordance with the 2014 Bethesda system]. However, the following participant may participate in this study; Atypical Squamous Cells of Undetermined Significance (ASC-US) and negative by high-risk Human Papillomavirus (HPV) test. And furthermore, regarding the participant with negative cervical cytology result conducted within 1 year, she may participate in this study without additional test.
13. The participant has a malignant tumor or a history of a malignant tumor within 5 years.
14. The participant has clinically significant cardiovascular disease or uncontrollable hypertension.
15. The participant is inappropriate for participation in this study based on 12-lead ECG findings, as determined by the investigator or subinvestigator.
16. The participant has active liver disease or jaundice, or has Alanine aminotransferase (ALT), Aspartate aminotransferase (AST) or total bilirubin > 1.5 times the upper limit of normal in the clinical laboratory tests.
17. The participant has previous or current history of diseases considered to be inappropriate for participation in this study, including severe hepatic impairment, jaundice, renal impairment, cardiovascular disease, endocrine system disease, metabolic disorder, pulmonary disease, gastrointestinal disease, neural disease, urological disease, immune disease, or mental disorder (especially depression-like symptoms) or suicide attempt resulting from a mental disorder.
18. The participant has a previous or current history of hypersensitivity to GnRH analogues, or has a previous or current history of severe hypersensitivity to other drugs.
19. The participant is pregnant, lactating, or intending to become pregnant or to donate ova between the signing date of informed consent and 1 month after the end of the study.

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 335 (Actual)
Dates: Start 2019-05-08 (Actual); Primary Completion 2020-06-12 (Actual); Study Completion 2020-09-28 (Actual)

PRIMARY OUTCOMES:
Change of maximum Visual Analogue Scale (VAS) score for endometriosis associated pelvic pain | Baseline and the last 28 days of treatment period
  Pelvic pain will be assessed using the VAS (0 - 100) as pain evaluation scale

SECONDARY OUTCOMES:
Change of mean VAS score for endometriosis associated pelvic pain | Baseline and the last 28 days of treatment period
  Pelvic pain will be assessed using the VAS (0 - 100) as pain evaluation scale
VAS score for endometriosis associated pelvic pain | Up to Week 24
  Pelvic pain will be assessed using the VAS (0 - 100) as pain evaluation scale
Change of VAS score for endometriosis associated pelvic pain | Baseline and up to Week 24
  Pelvic pain will be assessed using the VAS (0 - 100) as pain evaluation scale
VAS score for menstrual pain | Up to Week 24
  Menstrual pain will be assessed using the VAS (0 - 100) as pain evaluation scale
Change of VAS score for menstrual pain | Baseline and up to Week 24
  Menstrual pain will be assessed using the VAS (0 - 100) as pain evaluation scale
VAS score for endometriosis associated pelvic pain outside the menstruation period | Up to Week 24
  Pelvic pain outside the menstruation period will be assessed using the VAS (0 - 100) as pain evaluation scale
Change of VAS score for endometriosis associated pelvic pain outside the menstruation period | Baseline and up to Week 24
  Pelvic pain outside the menstruation period will be assessed using the VAS (0 - 100) as pain evaluation scale
VAS score for dyspareunia | Up to Week 24
  Dyspareunia will be assessed using the VAS (0 - 100) as pain evaluation scale
Change of VAS score for dyspareunia | Baseline and up to Week 24
  Dyspareunia will be assessed using the VAS (0 - 100) as pain evaluation scale
Adverse event | Up to Week 28
Bone mineral density | Up to Week 24
Serum concentrations of NTx (N-telopeptide) | Up to Week 24
Serum concentrations of BAP (Bone alkaline phosphatase) | Up to Week 24
Period from the last dose of study drug to return of menstrual cycles | From Week 24 to Week 28

CONTACTS AND LOCATIONS:
Locations (41):
- Japan (41):
  - Chubu Rosai Hospital, Aichi
  - Meitetsu Hospital, Aichi
  - Aiiku Ladies Clinic, Chiba
  - Chiba Aoba Municipal Hospital, Chiba
  - Tokyo Bay Urayasu Ichikawa Medical Center, Chiba
  - Tsujinaka Hospital Kashiwanoha, Chiba
  - Fujito Clinic, Hiroshima
  - Hashimoto Clinic, Hokkaido
  - Tokeidai Memorial Hospital, Hokkaido
  - Yoshio Obstetrics Gynecology Hospital, Hokkaido
  - Shinsuma Hospital, Hyōgo
  - Kagawa Prefectural Central Hospital, Kagawa
  - Takamatsu Red Cross Hospital, Kagawa
  - Fujisawa City Hospital, Kanagawa
  - Rinkan Clinic, Kanagawa
  - Second Kawasaki Saiwai Clinic, Kanagawa
  - Tawada Ladies Clinic, Kanagawa
  - Japanese Red Cross Kumamoto Hospital, Kumamoto
  - Kurashiki Medical Clinic, Okayama
  - Chayamachi Ladies Clinic, Osaka
  - Hayakawa Clinic, Osaka
  - Minami-Morimachi Ladies Clinic, Osaka
  - Nomura Clinic Nanba, Osaka
  - Rikako Ladies Clinic, Osaka
  - Tanabe Ladies Clinic, Osaka
  - Yoshimura Ladies Clinic, Osaka
  - Dantsuka Clinic, Saitama
  - Kashiwazaki Ladies Clinic, Saitama
  - Maruyama Memorial General Hospital, Saitama
  - Kusatsu General Hospital, Shiga
  - Akasaka-Mitsuke Miyazaki Clinic, Tokyo
  - Ginza Yoshida Hospital, Tokyo
  - Hamada Hospital, Tokyo
  - Ikebukuro Metroporitan Clinic, Tokyo
  - NS Clinic, Tokyo
  - Sei Women's Clinic, Tokyo
  - Seijo Kinoshita Hospital, Tokyo
  - Shimamura Memorial Hospital, Tokyo
  - Toranomon Women's Clinic, Tokyo
  - Yokokura Clinic, Tokyo
  - Yukawa Women's Clinic, Tokyo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Harada T, Osuga Y, Suzuki Y, Fujisawa M, Fukui M, Kitawaki J. Relugolix, an oral gonadotropin-releasing hormone receptor antagonist, reduces endometriosis-associated pain compared with leuprorelin in Japanese women: a phase 3, randomized, double-blind, noninferiority study. Fertil Steril. 2022 Mar;117(3):583-592. doi: 10.1016/j.fertnstert.2021.11.013. Epub 2021 Dec 8. PMID 34895700